CLINICAL TRIAL: NCT01397877
Title: Phase 2 Multicenter Study to Assess the Safety and Efficacy of BKM120 as Monotherapy in Treatment of Initial or Recurrent Metastatic Endometrial Cancer After 1st Line Therapy in Patients Who Cannot Undergo Local Surgery and/or Radiotherapy
Brief Title: GINECO-EN102b - BKM120 as Monotherapy in the Treatment of Initial or Recurrent Metastatic Endometrial Cancer
Acronym: ENDOPIK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDOPIK
Record Dates: First submitted 2011-07-18; First posted 2011-07-20 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; BKM; monotherapy; metastatic; initial treatment
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm Metastasis | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stratum 1 (Experimental): Patients with low grade disease (grade 1 or 2) with positive or negative mutational status
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — per os, 60mg/j, until progression or unacceptable toxicity

SUMMARY:
This study is to determine the clinical efficacy of BKM120 as monotherapy in the treatment of initial or recurrent metastatic endometrial cancer after first line radio chemotherapy.

Clinical efficacy will be determined by the non-progression rate at 3 or 2 months depending on the group of patients. The primary endpoint is the non-progression rate at 3 months (12 weeks) for the patient group whose disease is painless (low grade tumor = stratum 1) and the non-progression rate at 2 months (8 weeks) for the group of patients with an aggressive disease (high grade tumor = stratum 2).

Disease progression is defined by the RECIST 1.1 criteria

ELIGIBILITY:
Inclusion Criteria:

* Female ≥ 18 years
* ECOG ≤ 2
* Histologically confirmed endometrial cancer
* Not eligible for exclusive curative treatment by surgery and/or radiotherapy
* Initial metastatic endometrial cancer not treated with chemotherapy or radiotherapy prior to inclusion OR
* Recurrent endometrial cancer previously treated with adjuvant CT and RT, presenting with a disease-free interval of at least 12 months
* Presence of one or more measurable lesion(s) outside the irradiated areas
* Availability at inclusion of samples of tumor tissue (a block or at least 20 unstained slides) for tumor sub-classification and for routine molecular analysis
* Satisfactory biological functions: PNN ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, hemoglobin ≥ 9.0 g/dL, INR ≤ 2, standard normal values for potassium, calcium and magnesium, serum creatinine ≤ 1.5 x ULN or creatinine clearance > 50 mL/min, ALT and AST within normal range (or ≤ 3.0 x ULN if liver metastases present), Alkaline phosphatase ≤ 2.5 x ULN, serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert Syndrome), fasting glycemia ≤ 120 mg/dL or ≤ 6.7 mmol/L
* Life expectancy 3 months
* Post menopausal woman with at least 12 months of natural (spontaneous) amenorrhea
* Negative serum pregnancy test ≤ 72 hours prior to initiating treatment for woman of child-bearing potential
* Consent form signed before any procedure performed

Exclusion Criteria:

* Previous treatment with PI3K inhibitors and/or mTOR
* Presence of symptomatic CNS metastases. Patient must have completed any prior treatment for CNS metastases ≥ 28 days and, if on corticosteroid therapy, should be receiving a stable low dose
* Concomitant presence or history of another malignant tumor in the past 3 years prior to inclusion (except spinocellular or cutaneous basal cell epithelioma or non-melanomatous skin cancer treated successfully)
* Suffering from mood disorders based on an evaluation by the investigator or a psychiatrist OR with a given score according to the PHQ-9 or GAD-7 mood evaluation scale (cf protocol)
* Concomitant administration of another approved or investigational anticancer agent
* Pelvic and/or para-aortic radiotherapy within ≤ 28 days prior to inclusion or persistent side effects from this treatment on implementation of the selection procedures
* Major surgery during the 28 days prior to starting investigational drug or persistent side effects from surgery
* Uncontrolled diabetes (HbA1c > 8 %)
* Presence of an active heart disease, especially: LVEF < 50 % determined by MUGA or ECHO, QTc > 480 msec on ECG recorded during selection (with QTcF formula), angina warranting the administration of anti-angina treatment, ventricular arrhythmia except for benign premature ventricular contractions, supraventricular and nodal arrhythmias warranting a pacemaker or not controlled by a treatment, conduction anomalies warranting a pacemaker, valvular disease with documented involvement of cardiac function, symptomatic pericarditis
* History of heart disease
* Currently receiving treatment to prolong QT interval accompanied by a known risk of triggering wave burst arrhythmia. Impossible to stop treatment or to replace it before starting study medication
* GI dysfunction or disease that could significantly interfere with absorption of BKM120
* Chronic treatment with corticosteroids or other immunosuppressants
* Any other severe and/or uncontrolled concomitant disease, which is likely to contraindicate the patient's participation
* Known treatment non-compliance
* Currently receiving treatment known to be inhibitors or moderate and strong inducers of isoenzyme CYP3A. Impossible to stop this treatment or to replace it with a different treatment before starting the study product
* Severe pneumonitis
* Grade ≥ 3 biological anomalies
* Known history of HIV infection
* Pregnant woman or nursing mother

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Clinical Efficacy | 3 months
  To determine the clinical efficacy of BKM120 as monotherapy in the treatment of initial or recurrent metastatic endometrial cancer after first line radio chemotherapy.

SECONDARY OUTCOMES:
Safety according to CTCAE v4.0 criteria and mood questionnaires : PHQ-9 and GAD-7 | Patient will be followed for the duration of the study, an expected average of 75 days
  To assess patient safety and the tolerance of BKM120 administered as monotherapy at the daily dose of 100 mg.
Efficacy: PFS | 6 months
  To evaluate progression-free survival
Efficacy: ORR | Patient will be followed for the duration of the study, an expected average of 75 days
  To evaluate the objective response rate according to RECIST 1.1
Efficacy: overall survival | Patients will be followed for an expected average of 1 year and 75 days
  To evaluate overall survival.
Efficacy: duration of response | Patients will be followed for an expected average of 1 year and 75 days
  To evaluate the duration of the response. For patients in complete remission, the duration of the response will be calculated from the day on which a complete response is determined for the first time up to progression.
  For patients in partial remission, the duration of the response will be the overall response period calculated from the administration of the first treatment cycle up to the date of progression.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Ray-Coquard, MD, Principal Investigator — GINECO - Centre Léon Bérard
Locations (45):
- France (45):
  - Clinique Bonnefon, Alès
  - Centre Paul Papin, Angers
  - Institut Ste Catherine, Avignon
  - Hôpital jean Minjoz, Besançon
  - Centre Hospitalier de Blois, Blois
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - centre Francois baclesse, Caen
  - Centre jean Perrin, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - Centre Georges François leclerc, Dijon
  - Group Hospitalier Mutualiste de Grenoble, Grenoble
  - Hôpital Michallon - CHU Grenoble, Grenoble
  - CHD Les Oudairies, La Roche-sur-Yon
  - Hôpital André Mignot, Le Chesnay
  - Centre jean Bernard, Le Mans
  - Centre Oscar Lambret, Lille
  - CHU Dupuytren, Limoges
  - Centre Léon bérard, Lyon
  - Hôpital Prové Clairval, Marseille
  - institut Paoli Calmette, Marseille
  - CRLC Val d'Aurelle, Montpellier
  - Groupement de coopération sanitaire, Montpellier
  - Centre Alexis Vautrin, Nancy
  - Centre d'oncologie de Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - CHU Caremeau, Nîmes
  - Clinique Valdegour, Nîmes
  - Centre Hospitalier Régional, Orléans
  - Hopital Hotel Dieu, Paris
  - Hopital Tenon, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Frederic Joliot, Rouen
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Hôpital rené Huguenin, Saint-Cloud
  - ICO René Gauducheau, Saint-Herblain
  - Centre Etienne DOLET, Saint-Nazaire
  - Institut cancérologuie de la loire, Saint-Priest-en-Jarez
  - Hôpital Civil, Strasbourg
  - Centre Claudius Régaud, Toulouse
  - CHU Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif